CLINICAL TRIAL: NCT05505149
Title: Prognosis of Functionality in Cerebral Palsy: A Retrospektif Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abant Izzet Baysal University (Other)
Responsible Party: Principal Investigator, Seda AYAZ TAŞ, Assistant Professor, Abant Izzet Baysal University
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: BAIBU - SAT2
Record Dates: First submitted 2022-08-16; First posted 2022-08-17 (Actual); Last update posted 2022-08-17 (Actual); Status verified 2022-08

CONDITIONS: Cerebral Palsy
MeSH Terms: conditions — Cerebral Palsy | interventions — Physical Therapy Modalities

STUDY DESIGN:
Intervention Model Description: Preschool age group, school age group, adolescent age group
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 0 to 6 years old spastic cerebral palsy (Active Comparator): Children were individually included in the physiotherapy and rehabilitation program for 2 years, with 45 minutes each session, two days a week. All children's treatment program included targeted, personalized functional exercises according to neurodevelopmental treatment principles, and they were applied by the physiotherapists of the children in the rehabilitation centers.
  Interventions: Other: physiotherapy
- 7 to 12 years old spastic cerebral palsy (Active Comparator): Children were individually included in the physiotherapy and rehabilitation program for 2 years, with 45 minutes each session, two days a week. All children's treatment program included targeted, personalized functional exercises according to neurodevelopmental treatment principles, and they were applied by the physiotherapists of the children in the rehabilitation centers.
  Interventions: Other: physiotherapy
- 13 to 18 years old spastic cerebral palsy (Active Comparator): Children were individually included in the physiotherapy and rehabilitation program for 2 years, with 45 minutes each session, two days a week. All children's treatment program included targeted, personalized functional exercises according to neurodevelopmental treatment principles, and they were applied by the physiotherapists of the children in the rehabilitation centers.
  Interventions: Other: physiotherapy

INTERVENTIONS:
Other: physiotherapy — Children were individually included in the physiotherapy and rehabilitation program for 2 years, with 45 minutes each session, two days a week. All children's treatment program included targeted, personalized functional exercises according to neurodevelopmental treatment principles, and they were applied by the physiotherapists of the children in the rehabilitation centers.

SUMMARY:
To purpose of this study is ;to evaluate prognosis of functionality in children with Cerebral Palsy in different age groups (preschool, school age and adolescence) and predict the progression of motor function according to different functional classification systems in children with CP over a 2 year period.

DETAILED DESCRIPTION:
Cerebral Palsy (CP) is defined as 'a group of persistent, non-progressive, postural and movement disorders that occur in the developing fetal or infant brain, causing activity limitation'. The European Cerebral Palsy Monitoring Group has divided CP into 3 classes as spastic, dyskinetic and ataxic types. Spastic type is divided into two as unilateral spastic type SP, where one half of the body is affected, and bilateral spastic type SP, where both halves of the body are affected. Researchers and clinicians typically group individuals with CP using descriptive classification systems according to the types of tone disorders, the distribution of motor deficits, or the level of independence. However, motor disorders in children with CP are often accompanied by sensory, perception, cognitive, communication, behavior and secondary musculoskeletal problems and epilepsy. In addition to impaired muscle tone, postural control and synergistic muscle activation in both proximal and distal body parts, muscle and joint contractures are observed as a result of muscle weakness, decreased exercise tolerance and limitation in functional activities. Since CP is an umbrella term that includes developmental problems in addition to motor disorders, many developmental areas should be evaluated. According to the World Health Organization's International Classification of Functioning, Disability and Health, the health status of the individual; should be evaluated in a holistic perspective, which includes the definition and evaluation of functions such as eating, drinking, dexterity, communication and mobility. The functional status of children with CP in different developmental areas is determined by developmental area-specific classification systems. The classification system is used to classify and categorize. Functional classifications in CP are used to facilitate communication between clinicians, to create homogeneous groups in clinical studies, and to customize the treatment and follow-up of the patient according to the individual. Determining the current functional status of children with CP with classification systems contributes to making predictions about the quality of life and functional status of the child and family. In addition, predictions about changes in gross motor functions of children with CP are helpful in developing programs to prepare children for adolescence and adulthood. Because the stability of the system that classifies gross motor skills is still unclear, especially in adolescence. Determining the stability of the system that classifies gross motor skills in children with CP during their transition to adulthood will be critical in determining the prognosis of motor functions in adolescence. In children with CP, hand functions are restricted at different levels according to the extremity involvement affected by spasticity. Since the lower extremity involvement of the child with spastic diparetic CP is more, bimanual hand skills can be better classified. A child with quadriparetic CP may have limited hand skills since all four extremities are involved. For this reason, we think that determining the stability and progression of the manual skills classification systems in the rehabilitation process is important in terms of evaluating the success of the rehabilitation and the development of the child's participation in activities of daily living, eating and drinking functions.

Cognitive disorders may accompany motor skills disorders in children with CP. In the study of Unes et al., which included 225 children with CP, it was reported that cognitive skills were impaired in 45% of children, and this could negatively affect their communication skills. In the literature, gross motor functions of individuals with CP 'Gross Motor Function Classification System (GMFCS)', hand skills 'Manual Ability Classification System (MACS)', communication skills 'Communication Function Classification System (CFCS)', eating and drinking skills 'Eating and Drinking Ability Classification System (EDACS)'.

To reveal the functional status of children with CP in different age groups (preschool, school age and adolescence); We think that it will evaluate the child holistically, provide information about the future functional level of the child, and help shape the existing treatment programs according to different age groups.

The design of this study is a retrospective cohort study. Children with spastic type Cerebral Palsy between the ages of 0 and 18 who received physiotherapy at Ereğli Private Gökkuşağı Special Education and Rehabilitation Center and Düzce Private Gökkuşağı Special Education and Rehabilitation Center were included. Functionality of 108 children with spastic type Cerebral Palsy was evaluated by the researcher (S.A.T) over two years. The children participated in the physiotherapy program, during 45 minutes two times for a week over two years. All children's treatment program included targeted, personalized functional exercises according to neurodevelopmental treatment principles, and they were applied by the physiotherapists of the children in the rehabilitation centers. The children were divided into 3 groups according to their age: 0-6 (preschool), 7-12 (school age), 13-18 (adolescent). The first evaluation was made in February 2020 and the last evaluation was made twice, in February 2022. After the demographic characteristics of the children (age, gender, CP type) were taken, their functionalities were 'Gross Motor Function Classification System (KMFSS)', 'Manual Ability Classification System (MACS)', 'Communication Function Classification System (CFCS)' and 'Eating and Drinking Ability Classification'. System (EDACS)' was classified.

The eligibility criteria were as follows: (1) being aged between 0-18 years old, (2) being diagnosed with spastic type CP. The exclusion criteria were as follows: (1) having botulinum toxin injection; (2) having orthopedic surgery; (3) having epileptic seizures.

The sample size and power calculation were performed using the G*Power 3.1 power analysis program. The calculations were based on an odds ratio of 1.9 (calculated from the pilot study), an alpha level of 0.05, and the desired power of 80%. These parameters generate a necessary sample size of at least 101. To allow for dropouts, 125 children with CP were invited to study.

Statistical Package for Social Science (SPSS) version 21.0 for Windows software (SPSS, Inc., Chicago, IL, USA) was used for all statistical analyses. Before the statistical analysis, the Kolmogorov-Smirnov test was used to assess the data's distribution. Descriptive statistics, including frequency, the percentage for nominal variables, and mean and standard deviation for continuous variables were calculated. "Binary Logistic Regression Analysis" was used in the analysis of the model testing whether children with CP's age, sex, type of CP, Gross Motor Function Classification System level, Manual Ability Classification System level, Communication Function Classification System level, Eating and Drinking Ability Classification System level predict improvement in Gross Motor Function Classification System level (yes or no) after physiotherapy. The Enter method was used, and the Hosmer-Lemeshow (H-L) test was done for assessing the goodness of fit of the fitted logistic regression model. The results were evaluated by considering the model fit statistics and parameter significance and the significance level was set at p<0.05.

ELIGIBILITY:
Inclusion Criteria:

* being aged between 0-18 years old,
* being diagnosed with spastic type CP.

Exclusion Criteria:

* having botulinum toxin injection
* having orthopedic surgery
* having epileptic seizures.

Ages: 6 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 108 (Actual)
Dates: Start 2020-02-01 (Actual); Primary Completion 2022-02-01 (Actual); Study Completion 2022-02-01 (Actual)

PRIMARY OUTCOMES:
Gross Motor Function Classification System (GMFCS) | two years
  The GMFCS is a system that classifies the gross motor functions of the child with CP. This system includes five levels: 1 (most independent) to level 5 (fully dependent).

SECONDARY OUTCOMES:
Manual Ability Classification System (MACS) | two years
  The MACS is a classification system developed to classify manual skills for children with CP aged 4-18. This system includes five levels: 1 (most independent) to level 5 (fully dependent). In this study, Mini MACS was also used to classify the hand skills of children aged 0-4.
Communication Function Classification System (CFCS) | two years
  The CFCS is a valid and reliable system that classifies the communication skills of children with CP at the level of activity and participation. This system includes five levels: 1 (most independent) to level 5 (fully dependent).
Eating and Drinking Ability Classification System (EDACS) | two years
  The EDACS is used for classify the eating and drinking skills of children with CP. This system includes five levels: 1 (most independent) to level 5 (fully dependent)

CONTACTS AND LOCATIONS:
Overall Officials: Seda AYAZ TAŞ, Principal Investigator — Abant Izzet Baysal University
Locations (1):
- BAIBU, Bolu, Turkey (Türkiye)